CLINICAL TRIAL: NCT03388853
Title: Efficacy and Safety Study of Acetylcysteine/Doxofylline 1200/400 mg Effervescent Tablet in the Treatment of Moderate-Severe Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Efficacy and Safety Study of Acetylcysteine/Doxofylline 1200/400 mg Effervescent Tablet in the Treatment of Moderate-Severe COPD.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Neutec Ar-Ge San ve Tic A.Ş (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NEU-06.15
Record Dates: First submitted 2017-12-12; First posted 2018-01-03 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2017-12

CONDITIONS: COPD
Keywords: Acetylcysteine/Doxofylline; Acetylcysteine; Doxofylline; Effervescent Tablet; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Acetylcysteine; doxofylline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acetylcysteine/Doxofylline (Experimental): Acetylcysteine/Doxofylline 1200/400 mg Effervescent Tablet once daily for four weeks.
  Interventions: Drug: Acetylcysteine/Doxofylline
- Placebo (Placebo Comparator): Placebo once daily for four weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Acetylcysteine/Doxofylline — Acetylcysteine/Doxofylline 1200/400 mg Effervescent Tablet once daily for four weeks.
  Other Names: Mucofix 1200/400 mg Effervescent Tablet
  Arms: Acetylcysteine/Doxofylline
Other: Placebo — Placebo once daily for four weeks.
  Arms: Placebo

SUMMARY:
The objective is to assess efficacy and safety of Acetylcysteine/Doxofylline 1200/400 mg Effervescent Tablet once daily treatment besides standard/usual treatment, as compared with placebo once daily in patients with stable moderate to severe COPD.

DETAILED DESCRIPTION:
The objective is to assess efficacy and safety of Acetylcysteine/Doxofylline 1200/400 mg Effervescent Tablet once daily treatment besides standard/usual treatment, as compared with placebo once daily in patients with stable moderate to severe COPD.

Patients who met all inclusion criteria will be randomized to receive double-blind treatment with Acetylcysteine/Doxofylline 1200/400 mg Effervescent Tablet once daily (n = 35) or placebo (n = 35) once daily for 4 weeks.

Patients will be evaluated at 2 consecutive visits: screening & treatment visit (first visit) and after treatment visit (second visit).

Spirometric measurements will be performed at pre-treatment during the first visit and post-treatment at two different time points (23 hr + 15 min and 23 hr + 45 min) during the second visit. The average of the values at 23 hr 15 min and 23 hr 45 min during the second visit will be defined as trough value.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥40 years with moderate-severe COPD diagnosis according to the GOLD and on a therapeutic regimen for COPD for a year
* Patients with post-bronchodilator FEV1/FVC ratio <0.70
* Patients with post-bronchodilator FEV1≥30% and <80% of predicted normal value.
* Current smokers or ex-smokers with a smoking history of at least 10 pack-years
* Patients who have no exacerbation within last 4 weeks
* Females patients with childbearing potential using effective birth control method
* Patients who have a capability of communicate with investigator
* Patients who accept to comply with the requirements of the protocol
* Patients who signed written informed consent prior to participation

Exclusion Criteria:

* History of hypersensitivity to drugs contain Acetylcysteine or Doxofylline or other mucolitics or xanthines
* Patients who use mucolitic and/or xantines derivatives or ephedrine routinely.
* Patients who use CPAP (continous positive airway measure), BiPAP (bilevel continous positive airway measure) or mechanical ventilation
* History of chronic respiratory diseases except COPD.
* Patients who had COPD exacerbation or lower respiratory track infections that required antibiotic, oral or parenteral corticosteroid treatment within 4 weeks prior to first visit.
* Patients who have a history of myocardial infarction, hearth failure, acute ischemic coroner disease or severe cardiac arrhythmia requiring treatment within least 6 weeks.
* History of significant or uncontrolled disease or operation that may preclude participant from participating in the study
* Patients who have lung cancer
* Patients who had lung volume reduction operation
* Women patients who are pregnant or nursing
* History of allergic rhinitis or atopy
* Patients who have known serious prostatic hypertrophy or narrow-angle glaucoma requiring drug therapy
* History of alcohol abuse.

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2019-12-21 (Actual); Study Completion 2019-12-21 (Actual)

PRIMARY OUTCOMES:
Mean changes in Breathlessness, Cough, and Sputum Scale (BCSS) score from baseline | 4 weeks

SECONDARY OUTCOMES:
Mean changes in Clinical COPD Questionnaire (CCQ) score from baseline | 4 weeks
Mean changes in Modified Medical Research Council dyspnea scale (mMRC) from baseline | 4 weeks
Mean changes in FEV1 from baseline | 4 weeks
Mean changes in FVC from baseline | 4 weeks
Mean changes in serum C-reactive protein (CRP) concentration from baseline | 4 weeks
Evaluation of safety of study drug | 4 weeks
  Number of participants with treatment-related adverse events and/or abnormal laboratory values.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Cukurova University Faculty of Medicine, Chest Diseases Department, Adana
  - Health Sciences University, Sureyyapasa Chest Diseases and Thoracic Surgery Training and Research Hospital, Istanbul